CLINICAL TRIAL: NCT03343262
Title: Mechanisms Underlying the Regulation of Impaired Glucose Tolerance by Auricular Concha Electro-acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Peijing Rong, The deputy director of Institute of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChinaACMS-4
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ta-VNS "yidan-pi" (Experimental): Device:ta-VNS & Electro-acupuncture("yidan-pi" auricular acupoints):2 times per day,2 days per week for 12 weeks
  Interventions: Device: ta-VNS; Other: Electro-acupuncture
- ta-VNS "jian" (Placebo Comparator): Device:ta-VNS & Electro-acupuncture("jian" auricular acupoints):2 times per day,2 days per week for 12 weeks
  Interventions: Other: Electro-acupuncture

INTERVENTIONS:
Device: ta-VNS — The transcutaneous vagus nerve stimulation (taVNS) at auricular concha is a typical representative of TCM modernization. The taVNS regulates the autonomic nervous system, which shows a good therapeutic effect for the treatment of IGT.
  Other Names: transcutaneous vagus nerve stimulation
  Arms: ta-VNS "yidan-pi"
Other: Electro-acupuncture — one of the most common acupuncture methods, selecting acupoints based on traditional Chinese medicine theory. It exerts the function to regulate qi and blood circulation and balance Yang and Yin energy inside body.

SUMMARY:
Impaired Glucose Tolerance (IGT) is an abnormal metabolic state following glucose metabolic steady state but prior to diabetes. IGT is an important stage during the progression of diabetes, with an underlying mechanism of insulin resistance and pancreatic β cell dysfunction. IGT is one of the diseases that shows significant beneficial response to acupuncture treatment. Original findings from the investigators'laboratory show that transcutaneous auricular vagus nerve stimulation (taVNS) which is innervated by vagus nerve, would enhance the activity of pancreatic β cells, promote the secretion of insulin, upregulate the expression of insulin receptors in central as well as peripheral tissues, thus to improve glycometabolism. In this study, the investigators would further illuminate the mechanism of taVNS at "yidan-pi" auricular acupoints on the regulation of glucose metabolism, its improvement of the IGT state in rat model, as well as its regulation effect on insulin receptor expression and insulin resistance, and systematically illustrate the clinical effective of this treatment on IGT, with emphasize on its influence on the concentrations of glucose and HbA1c, and thus provide an effective proposal for clinical acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* ages between 20 and 70
* fasting plasma-glucose(FPG) less than 7 mmol/L, or 2h p-glucose 7.8-11.1 mmol/L
* anti-diabetic medication of any kind
* able to provide informed consent

Exclusion Criteria:

* comorbidities that would prohibit participation in study procedures, including cardiovascular disease, hematological system disease or psychosis
* females of childbearing potential who were pregnant, breast-feeding
* infection within the 1 month
* known or suspected abuse of alcohol or narcotics

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
FPG | Baseline and 6 week, 12 weeks
  The fasting plasma glucose (FPG) is used to diagnose diabetes. IGT can be diagnosed base on FPG less than 7.0 mmol/L.
OGGT | Baseline and 6 week, 12 weeks
  The 2-hour plasma glucose after a 75-g oral glucose tolerance test (OGTT) is used to diagnose diabetes. IGT can be diagnosed base on 2-hour plasma Glucose between 7.8 and 11.1 mmol/L.

SECONDARY OUTCOMES:
BMI | Baseline and 12 weeks
  The body mass index are used to diagnose Obesity. Weight and height will be combined to report BMI in kg/m^2
A1C | Baseline and 6 week,baseline and 12 weeks
  The hemoglobin A1C (A1C) is a diagnostic test for diabetes. Diabetes can be diagnosed base on A1C more than 6.5%.

OTHER OUTCOMES:
pulse | Baseline and 12 weeks
  Normal pulse should be more than 60 per minute, or less than 100 per minute.
respiration | Baseline and 12 weeks
  Normal respiration should be more than 16 times, or less than 20 times.
blood pressure | Baseline and 12 weeks
  The systolic pressure should be no more than 139 mmHG, and the diastolic pressure should be no less than 89 mmHg.
body temperature | Baseline and 12 weeks
  Normal temperature should be more than 36 C, or less than 37 C.

CONTACTS AND LOCATIONS:
Overall Officials: Peijing Rong, doctor, Study Director — Institute of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided